CLINICAL TRIAL: NCT03458650
Title: A Single-center, Randomized, Double-blinded and Placebo-controlled Clinical Study in Healthy Chinese Subjects to Evaluate the Pharmacokinetics, Safety and Tolerability of LXI-15028 After Receiving Escalating Single Oral Doses of LXI-15028 at 50 mg, 100 mg and 200 mg and Multiple Oral Doses of LXI-15028 at 100 mg
Brief Title: A Phase I Study of LuoXin Innovate (LXI-15028) in Healthy Chinese Subjects to Evaluate the Pharmacokinetics, Safety and Tolerability.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Luoxin Pharmaceutical Group Stock Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NE821605
Record Dates: First submitted 2018-01-25; First posted 2018-03-08 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LXI-15028 50 mg (Experimental): For 50 mg dose groups, each is planned to enroll 12 healthy subjects (investigational drug :placebo=10:2), half males and half females. Five subjects of each gender will receive LXI-15028, while 1 subject of each gender will receive placebo
  Interventions: Drug: LXI-15028 50mg; Drug: Placebo
- LXI-15028 100 mg (Experimental): 100 mg dose group plans to enroll 14 healthy subjects (investigational drug:placebo=10:4), half males and half females. Five subjects of each gender will receive LXI-15028, while 2 subjects of each gender will receive placebo. Intra-group randomization will be implemented in each dose group; each subject will receive either LXI-15028 or placebo.
  Interventions: Drug: LXI-15028 100mg; Drug: Placebo
- LXI-15028 200 mg (Experimental): 200 mg dose groups, each is planned to enroll 12 healthy subjects (investigational drug :placebo=10:2), half males and half females. Five subjects of each gender will receive LXI-15028, while 1 subject of each gender will receive placebo
  Interventions: Drug: LXI-15028 200mg; Drug: Placebo

INTERVENTIONS:
Drug: LXI-15028 50mg — In escalated single-dose study, the subjects in each dose group will receive single oral dose of 50 mg LXI-15028 tablet or 1 matching placebo tablet at fasted state,
  Arms: LXI-15028 50 mg
Drug: LXI-15028 100mg — 100 mg LXI-15028 tablet or matching placebo 1 tablet at fasted state, In multiple-dose study, the subjects who administered 100mg single dose will continuously receive oral 100 mg LXI-15028 tablet or 1 matching placebo tablet once daily (QD) for 10 times.
  Arms: LXI-15028 100 mg
Drug: LXI-15028 200mg — single oral dose 2 100 mg LXI-15028 tablets or 2 matching placebo tablets at fasted state
  Arms: LXI-15028 200 mg
Drug: Placebo — matching placebo tablets

SUMMARY:
"This study is a single-center, randomized, double-blinded and placebo-controlled trial designed not only to assess pharmacokinetics, safety and tolerability of LXI-15028 but also to evaluate the pharmacokinetic characteristics of main metabolite M1 in vivo in 38 healthy adult Chinese subjects after receiving escalating single oral doses of 50 mg, 100 mg and 200 mg and multiple oral doses of 100 mg of LXI-15028.

DETAILED DESCRIPTION:
This study includes 3 dose groups which are 50 mg (Group 1), 100 mg(Group 2) and 200 mg(Group 3) respectively. For 50 mg and 200 mg dose groups, each is planned to enroll 12 healthy subjects (investigational drug :placebo=10:2), half males and half females. Five subjects of each gender will receive LXI-15028, while 1 subject of each gender will receive placebo; 100 mg dose group plans to enroll 14 healthy subjects (investigational drug:placebo=10:4), half males and half females. Five subjects of each gender will receive LXI-15028, while 2 subjects of each gender will receive placebo. Intra-group randomization will be implemented in each dose group; each subject will receive either LXI-15028 or placebo.

This study includes 2 parts of single-dose and multiple-dose administration. The single-dose study will use gradually escalation dosing to evaluate the 3 doses of 50 mg, 100 mg and 200 mg. Within 4 days after each dose is administered, the investigators will assess the safety and tolerability data to decide whether to proceed with the next escalated single dose. Within 4 days of 200 mg single-dose administration, the investigators will assess the safety and tolerability data to decide whether to proceed with 100 mg multiple-dose study. Multiple-dose study will be investigated in 100 mg group only.

The study consists of screening period, treatment period and follow-up in each dose group. The treatment period in 50 mg and 200 mg dose groups include single-dose administration only. While the treatment period in 100 mg dose group includes both single-dose and multiple-dose administration. The subjects in 100 mg dose group will enter multiple-dose period following completing single-dose period.

In escalated single-dose study, the subjects in each dose group will receive single oral dose of 50 mg LXI-15028 tablet or 1 matching placebo tablet at fasted state, or 100 mg LXI-15028 tablet or matching placebo 1 tablet, or 2 100 mg LXI-15028 tablets or 2 matching placebo tablets. Blood samples will be collected before administration (0h), and 15 min (0.25h), 30 min (0.5h), 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h, 24h, 48h and 72h after administration. In multiple-dose study, the subjects will continuously receive oral 100 mg LXI-15028 tablet or 1 matching placebo tablet once daily (QD) for 10 times. Blood samples of trough concentration will be collected before the 8th to 10th administration (0h) in multiple-dose study. And blood samples will be collected at 15 min (0.25h), 30 min (0.5h), 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h, 24h, 48h and 72h after the 10th administration.

The collected blood samples will be processed to obtain plasma. Liquid Chromatographic(LC) /Mass Spectra(MS)/Mass Spectra (MS) method will be used to determine plasma concentrations of LXI-15028 and its major metabolite M1 in order to evaluate the pharmacokinetic characteristics of LXI-15028 and its metabolite M1 after oral administration of LXI-15028 tablet.

The safety will be assessed by physical examination, vital signs, ECG, laboratory examinations and adverse events in subjects receiving LXI-15028 tablet.

"

ELIGIBILITY:
Inclusion Criteria:

* The subjects should voluntarily participate in this trial and sign the informed consent form prior to conducting any trial-related procedures;
* Gender: male or female healthy subjects; Age: 18~45 years old (including 18 and 45 years old);
* The body weight should be equal or greater than 50.0 kg for male and 45.0 kg for female. Body weight index (BMI)= body weight (kg)/[height(m)×height(m)], should be within the range from 19 to 25 (including 19 and 25);
* In the past three years, no history or presence of cardiovascular, hepatic, renal, respiratory, hematological and lymphatic, endocrine, immunological, mental, neurological and gastrointestinal disease; no history of surgery;
* The subjects (including males and females) agree to use medically approved contraceptive methods during the trial period and within 3 months after the end of the trial in order to avoid pregnancy; medically approved contraceptive methods include intrauterine device, physical barrier (male condom, female condom), subcutaneous implant, sustained-release contraceptive, bilateral salpingectomy, bilateral tubal ligation, bilateral vas ligation, etc.;
* The subjects agree not to donate sperms (males) or ova (females) at least 7 days before the first dose, during the study and within 3 months after ending of this study.

Exclusion Criteria:

* The subjects with allergic constitution, for example those with bronchial asthma, allergic to food or pollen, allergic to two or more drugs or those with known history of allergy ; or the subjects with any serious adverse response to Proton Pump Inhibitor or P-CABs previously (e.g., omeprazole, rabeprazole, lansoprazole and TAK-481 ), or known allergy to penicillins or cephalosporins;
* The investigator determines that it may potentially affect absorption, distribution, metabolism or elimination of investigational drug (e.g. organ dysfunction);
* The subjects with a history of drug abuse or drug abuse screening positive;
* The subjects received any drugs (including prescription drugs, Over-The-Counter drugs, herbal medicines, etc.) within 1 month before the screening or are taking drugs, especially CYP3A inhibitor or inducer (see Appendix 1);
* The subjects with clinical significant physical examination abnormalities determined by investigator;
* Heart rate<50 beats/min or >100 beats/min or QTc interval prolonged (male QTcF≥430ms, female QTcF≥450ms) or QRS≥120 msec or other clinically significant ECG abnormalities; 7) The subjects with sitting blood pressure: systolic pressure <90mmHg or ≥ 140mmHg, diastolic pressure ≥90mmHg or <60mmHg, which shows clinical significant abnormalities determined by investigators
* The subjects with any biomarker value of Aspartate aminotransferase (AST),Alanine aminotransferase(ALT), Alkaline phosphatase(ALP),r-Glutamyl Transferase (r-GT), total bilirubin, creatinine above the upper limit of normal or with other clinical significant laboratory examination abnormalities judged by investigators
* The subjects with presence of one of the following infectious diseases;

  1. Virological determination indicates hepatitis B virus surface antigen (HBsAg) positive or anti-hepatitis C virus antibody positive;
  2. Acquired human immunodeficiency virus determination indicates infection; (anti-human immunodeficiency virus antibody positive)
  3. Treponema pallidum infection (anti-treponema pallidum-specific antibody positive).
* Currently smoking or quitting smoking less than 3 months before screening or tobacco screening positive;
* Chronical alcohol user within 5 years prior to screening, or alcohol consumption of more than 14 unit alcohol per week (1 unit alcohol equal to 360 mL beer, or 150 mL grape wine, or 45 mL wine of 40 degree) within 6 months prior to screening;
* Alcohol screening test positive or alcohol intake within 72 h prior to screening;
* Daily drinking a large amount (above 1000 mL) of tea, coffee, cola and/or caffeine-containing beverages within 6 months prior to screening;
* Taking xanthine-containing or caffeine-containing food or beverages (including chocolate, tea, coffee and cola, etc.) from 48 hours prior to screening;
* Taking grapefruit, lime, carambola or any food or beverages made from them within 7 days prior to screening;
* Female subjects with blood pregnancy test positive or during lactation
* Difficulty in blood sampling, or has relevant history, symptoms or signs of blood sampling difficulty;
* Transfusion treatment or blood donation or massive blood loss (exceeding 450 mL) judged by investigators within 3 months prior to screening;
* Participation in any other clinical study within 3 months prior to screening;
* Participation in the planning or execution of this study (e.g., the sponsor or staff in the site);
* Inappropriate to participate in this study for any reason according to the medical judgment of investigators.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2018-04-23 (Actual); Study Completion 2018-05-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter： Cmax | 72 h after receiving single oral dose
  The maximum plasma concentration (Cmax) after single dose LXI-15028
Pharmacokinetic parameter： Tmax | 72 h after receiving single oral dose
  The peak time (Tmax) after single dose LXI-15028
Pharmacokinetic parameter： T1/2 | 72 h after receiving single oral dose
  The elimination half-life T1/2 after single dose LXI-15028
Pharmacokinetic parameter： Kel | 72 h after receiving single oral dose
  The eliminate rate constant after single dose LXI-15028
Pharmacokinetic parameter：Mean Residence Time(MRT) | 72 h after receiving single oral dose
  The mean residence time after single dose LXI-15028
Pharmacokinetic parameter: Area Under plasma Concentration(AUC 0-24h) | 24h after receiving single oral dose
  The area under plasma concentration -time curve from 0 time ot 24 h after single dose LXI-15028
Pharmacokinetic parameter: AUC 0-last | 72h after receiving single oral dose
  The area under plasma concentration- time curve from 0 time to sampling time of the last measurable concentration after single dose LXI-15028
Pharmacokinetic parameter: AUC 0-inf | 72h after receiving single oral dose
  The area under plasma concentration-time curve from adminstration (0)to infinity after single dose LXI-15028
Pharmacokinetic parameter: Vd/F | 72h after receiving single oral dose
  The apparent volume of distribution after single dose LXI-15028
Pharmacokinetic parameter: Css min | predose at day 8, 9, and 10, 72 h after receiving last multiple oral doses
  The trough concentration at steady state(Css min) after multiple doses
Pharmacokinetic parameter: Css max | 72 h after receiving last multiple oral doses
  The peak concentration at steady state (Css max) after multiple doses
Pharmacokinetic parameter: Css av | 72 h after receiving last multiple oral doses
  The average concentration at steady state (Css, av)after multiple doses
Pharmacokinetic parameter: Tss max | 72 h after receiving last multiple oral doses
  The peak time after multiple doses
Pharmacokinetic parameter: Tss,1/2 | 72 h after receiving last multiple oral doses
  The steady-state clearance half-time after multiple doses
Pharmacokinetic parameter: CLss/F | 72 h after receiving last multiple oral doses
  Total body clearance after multiple doses
Pharmacokinetic parameter: coefficient of fluctuation (DF) | 72 h after receiving last multiple oral doses
  coefficient of fluctuation after multiple doses
Pharmacokinetic parameter: Area Under plasma Concentration at steady state (AUC ss) | 72 h after receiving last multiple oral doses
  The area under plasma concentration-time curve at steady state after multiple doses
Pharmacokinetic parameter: Rac | 72 h after receiving last multiple oral doses
  The accumulation coefficient after multiple doses
Physical examination value of single dose | Baseline to Day 4 after receiving single oral dose
  This measure is a composite. Evaluate safety and tolerability of single dose in Physical examination that should cover the head, eyes, ears, nose, throat, cardiovascular system, skin, musculoskeletal, respiratory system, digestive system, urinary system and nervous system and changes of each item from the baseline are summarized. The measurement results of each subject are summarized by different severity. All physical examination results during this trial will be listed in details.
Vital signs value of single dose | Up to 3weeks
  The measure is a composite.Evaluate safety and tolerability of single dose in Vital signs value that including blood pressure (Systolic blood pressure/Diastolic blood pressure), pulse, body temperature，each vital sign examination values at each evaluation time point and their changes relative to the baseline will be summarized. All vital sign results should be listed. The listed vital signs are compared with normal ranges to determine whether is abnormal. The examination results that are divided into higher than normal range, normal and lower than normal range will be summarized by number of cases (n) and percentage (%). The results of abnormalities(> or < normal range) are listed.
12-lead ECG value of single dose | Up to 3 weeks
  Evaluate safety and tolerability of single dose in 12-lead ECG value that including ventricular rate (beats/min), PR interval (ms), QRS (ms) , QT(ms),QTc (ms)， the examination results of each ECG parameters and their changes from baseline will be summarized at each time point. Meanwhile, all 12-lead ECG examination results will be listed in details.
Blood routine value of single dose | Baseline to Day 4 after receiving single oral dose
  Evaluate safety and tolerability of single dose in blood routine value that including White blood cells (WBC), red blood cells (RBC), hemoglobin (Hb), hematocrit (Hct), platelet, neutrophils, lymphocytes, monocytes, eosinophils, basophils, absolute neutrophil counts (ANC);and list all the result.
Urine routine value of single dose | Baseline to Day 4 after receiving single oral dose
  Evaluate safety and tolerability of single dose in urine routine value that including specific gravity, pH, proteins, ketone,occult blood; and list all the result.
Blood coagulation value of single dose | Baseline to Day 4 after receiving single oral dose
  Evaluate safety and tolerability of single dose in blood coagulation value that including International normalized ratio (INR), activated partial thromboplastin time (aPTT), prothrombin time (PT); and list all the result.
Blood biochemistry value of single dose | Baseline to Day 4 after receiving single oral dose
  Evaluate safety and tolerability of single dose in blood biochemistry value that including Cholesterol, total proteins, albumin, total bilirubin, Conjugated bilirubin, creatinine, creatine kinase (CPK), alkaline phosphatase (ALP), aspartate aminotransferase (AST), alanine aminotransferase (ALT), glutamyltransferase (γ-GT), magnesium, sodium, potassium, chlorine, total calcium, inorganic phosphorus, lactate dehydrogenase (LDH), glucose, uric acid, triglyceride (TG); and list all the result.
Adverse events of single dose | Up to 3 weeks
  The adverse events are encoded using MedDRA 20.1. According to system organ classification (SOC) and preferred term (PT), all TEAE, investigational drug-related TEAE, Serious Adverse Event, investigational drug-related SAE, and TEAE causing premature withdrawal from this study will be separately summarized by different dose groups, including number of subjects experiencing Adverse Event, percentage and number of AE cases. The summary results are sorted according to the ranking number of cases of all subjects experiencing AE. All AE and SAE are listed by different dose groups.
Physical examination value of multiple doses | Baseline to Day 21 after receiving the first dose
  The measure is a composite. Evaluate safety and tolerability of multiple doses in Physical examination that should cover the head, eyes, ears, nose, throat, cardiovascular system, skin, musculoskeletal, respiratory system, digestive system, urinary system and nervous system and changes of each item from the baseline are summarized. The measurement results of each subject are summarized by different severity. All physical examination results during this trial will be listed in details.
Vital signs value of multiple doses | Baseline to Day 21 after receiving the first dose
  The measure is a composite.Evaluate safety and tolerability of multiple doses in Vital signs value that including blood pressure(Systolic blood pressure/Diastolic blood pressure), pulse, body temperature.Each vital sign examination values at each evaluation time point and their changes relative to the baseline will be summarized. All vital sign results should be listed. The listed vital signs are compared with normal ranges to determine whether is abnormal. The examination results that are divided into higher than normal range, normal and lower than normal range will be summarized by number of cases (n) and percentage (%). The results of abnormalities(> or < normal range) are listed.
12-lead ECG value of multiple doses | :Baseline to Day 21 after receiving the first dose
  Evaluate safety and tolerability of multiple doses in 12-lead ECG value that including ventricular rate (beats/min) ，PR interval (ms)， QRS (ms) ,，QT(ms)， QT interval (QTc )(ms). The examination results of each ECG parameters and their changes from baseline will be summarized at each time point. Meanwhile, all 12-lead ECG examination results will be listed in details.
Blood routine value of multiple doses | Baseline to Day 21 after receiving the first dose
  Evaluate safety and tolerability of multiple doses in blood routine value that including White blood cells (WBC), red blood cells (RBC), hemoglobin (Hb), hematocrit (Hct), platelet, neutrophils, lymphocytes, monocytes, eosinophils, basophils, absolute neutrophil counts (ANC); and list all the result.
Urine routine value of multiple doses | Baseline to Day 21 after receiving the first dose
  Evaluate safety and tolerability of multiple doses in urine routine value that including specific gravity, potential of hydrogen (pH), proteins, ketone,occult blood; and list all the result.
Blood coagulation value of multiple doses | Baseline to Day 21 after receiving the first dose
  Evaluate safety and tolerability of multiple doses in blood coagulation value that including International normalized ratio (INR), activated partial thromboplastin time (aPTT), prothrombin time (PT);
Blood biochemistry value of multiple doses | Baseline to Day 21 after receiving the first dose
  Evaluate safety and tolerability of multiple doses in blood biochemistry value that including Cholesterol, total proteins, albumin, total bilirubin, Conjugated bilirubin, creatinine, creatine kinase (CPK), alkaline phosphatase (ALP), aspartate aminotransferase (AST), alanine aminotransferase (ALT), glutamyltransferase (γ-GT), magnesium, sodium, potassium, chlorine, total calcium, inorganic phosphorus, lactate dehydrogenase (LDH), glucose, uric acid, triglyceride (TG); and list all the result.
Adverse events of multiple doses | Up to 6 weeks
  The adverse events are encoded using MedDRA 20.1. According to system organ classification (SOC) and preferred term (PT), all treatment-emergent adverse event (TEAE), investigational drug-related TEAE, serious adverse event (SAE), investigational drug-related SAE, and TEAE causing premature withdrawal from this study will be separately summarized by different dose groups, including number of subjects experiencing AE, percentage and number of adverse event (AE) cases. The summary results are sorted according to the ranking number of cases of all subjects experiencing AE. All AE and SAE are listed by different dose groups.

SECONDARY OUTCOMES:
Pharmacokinetic parameter of major metabolite(M1): Cmax | 72 h after receiving single oral doses
  Major metabolite (M1) of LXI-15028 Plasma PK parameters of single doses: peak concentration Cmax
Pharmacokinetic parameter of major metabolite(M1): Tmax | 72 h after receiving single oral doses
  Major metabolite (M1) of LXI-15028 Plasma PK parameters of single doses: peak time Tmax
Pharmacokinetic parameter of major metabolite(M1): T1/2 | 72 h after receiving single oral doses
  Major metabolite (M1) of LXI-15028 Plasma PK parameters of single doses: elimination half-life T1/2
Pharmacokinetic parameter of major metabolite(M1): Kel | 72 h after receiving single oral dose
  Major metabolite (M1) of LXI-15028 Plasma PK parameters of single doses: eliminate rate constant
Pharmacokinetic parameter of major metabolite(M1): MRT | 72 h after receiving single oral dose
  Major metabolite (M1) of LXI-15028 Plasma PK parameters of single doses: mean residence time
Pharmacokinetic parameter of major metabolite(M1): AUC 0-24h | 24 h after receiving single oral dose
  Major metabolite (M1) of LXI-15028 Plasma PK parameters of single doses: area under plasma concentration-time curve from 0 time to 24 hours
Pharmacokinetic parameter of major metabolite(M1): AUC 0-last | 72 h after receiving single oral dose
  Major metabolite (M1) of LXI-15028 Plasma PK parameters of single doses: area under plasma concentration-time curve from 0 time to the last measurable concentration
Pharmacokinetic parameter of major metabolite(M1): AUC 0-inf | 72h after receiving single oral dose
  Major metabolite (M1) of LXI-15028 Plasma PK parameters of single doses: area under plasma concentration-time curve from 0 time to infinity
Pharmacokinetic parameter of major metabolite(M1): CL/F | 72h after receiving single oral dose
  Major metabolite (M1) of LXI-15028 Plasma PK parameters of single dose:apparent total clearance
Pharmacokinetic parameter of major metabolite(M1): Vd/F | 72h after receiving single oral dose
  Major metabolite (M1) of LXI-15028 Plasma PK parameters of single dose: apparent volume of distribution
Pharmacokinetic parameter of major metabolite(M1): Css, min | :predose at day 8, 9, and 10, 72 h after receiving last multiple oral doses
  Major metabolite (M1) of LXI-15028 Plasma PK parameters of multiple doses: trough concentration at steady state
Pharmacokinetic parameter of major metabolite(M1): Css, max | 72 h after receiving last multiple oral doses
  Major metabolite (M1) of LXI-15028 Plasma PK parameters of multiple doses:peak concentration at steady state
Pharmacokinetic parameter of major metabolite(M1): Css, av | 72 h after receiving last multiple oral doses
  Major metabolite (M1) of LXI-15028 Plasma PK parameters of multiple doses: average concentration at steady state
Pharmacokinetic parameter of major metabolite(M1): Tss, max | 72 h after receiving last multiple oral doses
  Major metabolite (M1) of LXI-15028 Plasma PK parameters of multiple doses: peak time
Pharmacokinetic parameter of major metabolite(M1): Vss/F | 72 h after receiving last multiple oral doses
  Major metabolite (M1) of LXI-15028 Plasma Pharmacokinetic parameters of multiple doses:apparent volume of distribution at steady state
Pharmacokinetic parameter of major metabolite(M1): tss,1/2 | 72 h after receiving last multiple oral doses
  Major metabolite (M1) of LXI-15028 Plasma Pharmacokinetic parameters of multiple doses:steady-state clearance half-life
Pharmacokinetic parameter of major metabolite(M1): CLss/F | 72 h after receiving last multiple oral doses
  Major metabolite (M1) of LXI-15028 Plasma Pharmacokinetic parameters of multiple doses:total body clearance
Pharmacokinetic parameter of major metabolite(M1): DF | 72 h after receiving last multiple oral doses
  Major metabolite (M1) of LXI-15028 Plasma Pharmacokinetic parameters of multiple doses: coefficient of fluctuation
Pharmacokinetic parameter of major metabolite(M1): AUCss | 72 h after receiving last multiple oral doses
  Major metabolite (M1) of LXI-15028 Plasma Pharmacokinetic parameters of multiple doses: area under plasma concentration-time curve at steady state
Pharmacokinetic parameter of major metabolite(M1): Rac | 72 h after receiving last multiple oral doses
  Major metabolite (M1) of LXI-15028 Plasma PK parameters of multiple doses: accumulation coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zhang, Doctor, Principal Investigator — Chief technician
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No